CLINICAL TRIAL: NCT03685435
Title: Preoperative Presence of Gastric Content in Non-fasting Patients - an Ultrasound Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Dahl, Professor 2, University Hospital, Akershus
Other Study IDs: 2018/1560
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Non-fasting Patients; Rapid Sequence Intubation; Anesthesia Intubation Complication
Keywords: Ultrasound; Gastric content; Non-fasting; Rapid Sequence Induction; Gastric volume

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-fasting patients: We will examine non-fasting patients using bedside ultrasound. First we examine the gaster in a supine position. Then we repeat the procedure in a right lateral position.
  Interventions: Other: Bedside ultrasound

INTERVENTIONS:
Other: Bedside ultrasound — Checking for gastric content using bedside ultrasound

SUMMARY:
Using bedside ultrasound, the investigators will examine gastric content in non-fasting patients assigned to rapid sequence intubation (RSI). The procedure will be done immediately before intubation. The percentage of non-fasting patients who actually have gastric content will be determined.

Identifying gastric content is critical because presence increases the risk of pulmonary aspiration during intubation.

DETAILED DESCRIPTION:
Quantitative gastric content will be registered by measuring the cross section area of antrum using bedside ultrasound. The area and the patients age will be applied to estimate gastric volume.

ELIGIBILITY:
Inclusion Criteria:

* adults scheduled for surgery
* Adults over 18 years old that are assigned to general anesthesia with rapid sequence intubation (RSI)

Exclusion Criteria:

* Body mass index over 40
* Pregnant women
* Patients earlier underwent gastric surgery
* Critically ill patients where spending time on ultrasound would cause a major disadvantage for the patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are assigned to rapid sequence intubation are considered non-fasting. Reasons for considering a patient non-fasting are among others: intake of food the last six hours, nausea, anxiety, preoperative intake of painkillers or reflux disease.
  The ultrasound method we are using, are only valid for this specific population.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-02-17 (Actual); Study Completion 2019-02-17 (Actual)

PRIMARY OUTCOMES:
High risk of aspiration | Immediately before intubation
  Detection of solids, or more than 1,5 mL/kg clear fluid in the gaster
Low risk of aspiration | Immediately before intubation
  Detection of empty stomach, or less than 1,5 mL/kg clear fluid in the gaster

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Dahl, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
We have not planned to share data with other researchers.